CLINICAL TRIAL: NCT04446819
Title: A Multicenter Prospective Phase III Clinical Study of Reducing Albumin-binding Paclitaxel Induced Peripheral Sensory and Motor Neurotoxicity of Upper Extremities With Compression Gloves (REMAINING)
Brief Title: Compression Gloves to Reduce Albumin-binding Paclitaxel Induced Peripheral Sensory and Motor Neurotoxicity (REMAINING)
Acronym: REMAINING
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Associate Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BUAY-20-01
Record Dates: First submitted 2020-06-18; First posted 2020-06-25 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Peripheral Neuropathy
Keywords: Paclitaxel; Compression gloves; Compression therapy; Neurotoxicity
MeSH Terms: conditions — Peripheral Nervous System Diseases; Neurotoxicity Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort (Other): Patients diagnosed with solid tumors who are about to received albumin-binding paclitaxel monotherapy are recruited. Dominant hands and non-dominant hands are treated with small-size compression gloves and suitable-size compression gloves, respectively, during the administration of albumin-binding paclitaxel.
  Interventions: Device: Compression gloves

INTERVENTIONS:
Device: Compression gloves — Patients wear small-size compression gloves (one or two size smaller than suitable size) for dominant hands and suitable-size compression gloves for non-dominant hands for 90 minutes during the administration of albumin-binding paclitaxel (start from 30 minutes before albumin-binding paclitaxel infusion).

SUMMARY:
Nanoparticle albumin-bound paclitaxel has greater efficacy and favorable safety profile than standard paclitaxel. However, rate of neuropathy caused by nanoparticle albumin-bound paclitaxel is higher than standard paclitaxel, and is one of its dose-limited toxicities. Previously, compression therapy by surgical gloves has shown effectiveness in preventing chemotherapy-induced neuropathy. We designed this multi-center prospective self-control phase III study to investigate the efficacy of compression gloves to reduce albumin-binding paclitaxel induced sensory and motor neurotoxicity of upper extremities.

ELIGIBILITY:
Inclusion Criteria:

* Patients are diagnosed with pathologically confirmed solid tumors.
* Patients are about to receive albumin-binding paclitaxel monotherapy (at least 4 cycles anticipated) by physicians' choice.
* Patients should have baseline Grade 0 peripheral sensory and motor neurotoxicity (NCI-CTCAE 5.0).
* Eastern Cooperative Oncology Group performance status ≤ 1.
* Biochemical tests within 7 days before inclusion should meet the following criteria:

  * Hemoglobin ≥ 90g/L, white blood cell count ≥ 3500/mm^3, neutrophil ≥ 1500/mm^3 and platelet ≥ 75000/mm^3 with no blood transfusion or hematopoietic colony-stimulating factors in the past 14 days.
  * Creatinine ≤ 1.5 times upper limit of normal (ULN).
  * Liver function: For patients without liver metastasis, alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) ≤ 1.5 times ULN, and total bilirubin ≤ 1.25 times ULN. For patients with liver metastasis, ALT, AST and ALP ≤ 5 times ULN and total bilirubin ≤ 1.5 times ULN.
* Life expectancy ≥ 12 weeks.
* No history of severe diseases in important organs including heart, lung, liver, and kidney.
* Willingness to sign a written informed consent.
* Willingness to adhere to dose and visit schedules.
* Women of child-bearing ages should be willing to take birth control methods during treatment and within 8 weeks after trial, and pregnancy test (blood or urine) within 14 days before inclusion should be negative (if positive, ultrasound should be performed to rule out pregnancy). Male patients should be willing to take birth control methods during treatment and within 8 weeks after trial or be sterilized by surgery .

Exclusion Criteria:

* Patients with uncontrolled and severe infection.
* Patients with meningeal metastasis, symptomatic brain metastasis, spinal cord compression, or new discovery of brain or pia mater diseases during screening. Patients who finish brain local control treatment, manifest stable symptoms and without brain hemorrhage in radiological screening can be included in the trial.
* Investigators decide the patient unsuitable for the trial.

Elimination Criteria:

* Patients have allergy to albumin-binding paclitaxel and are unable to finish 4 cycles of treatment.
* Patients are unable to finish 4 cycles of albumin-binding paclitaxel monotherapy due to intolerable toxicities even after twice dose reduction. If due to toxicity of peripheral neurotoxicity, evaluations should be performed and recorded for further case study.
* Patients are unable to finish 4 cycles of albumin-binding paclitaxel monotherapy because of change of regimen due to progression or death.
* Patients require to quit.
* Patients are found to have situations that are not suitable for the trial after inclusion.
* Patients' hands are unfit for the compression gloves used in the trial (too big or too small).
* Any situations that investigators believe necessary for patients to quit the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-07-12 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Differences in severe peripheral sensory neurotoxicity rates | 3 weeks after Cycle 4 administration and/or 1 day before Cycle 5 administration of albumin-binding paclitaxel (each cycle is 21 days).
  Differences in peripheral sensory neurotoxicity (NCI-CTCAE Grade 2-5) rates between dominant hands and non-dominant hands after 4 cycles of albumin-binding paclitaxel monotherapy.

SECONDARY OUTCOMES:
Differences in total peripheral sensory neurotoxicity rates | 3 weeks after Cycle 4 administration and/or 1 day before Cycle 5 administration of albumin-binding paclitaxel (each cycle is 21 days).
  Differences in total peripheral sensory neurotoxicity (NCI-CTCAE Grade 1-5) rates between dominant hands and non-dominant hands after 4 cycles of albumin-binding paclitaxel monotherapy.
Differences in severe peripheral motor neurotoxicity rates | 3 weeks after Cycle 4 administration and/or 1 day before Cycle 5 administration of albumin-binding paclitaxel (each cycle is 21 days).
  Differences in severe peripheral motor neurotoxicity (NCI-CTCAE Grade 2-5) rates between dominant hands and non-dominant hands after 4 cycles of albumin-binding paclitaxel monotherapy.
Differences in total peripheral motor neurotoxicity rates | 3 weeks after Cycle 4 administration and/or 1 day before Cycle 5 administration of albumin-binding paclitaxel (each cycle is 21 days).
  Differences in total peripheral motor neurotoxicity (NCI-CTCAE Grade 1-5) rates between dominant hands and non-dominant hands after 4 cycles of albumin-binding paclitaxel monotherapy.
Differences in peripheral neurotoxicity questionaire scores | 3 weeks after Cycle 4 administration and/or 1 day before Cycle 5 administration of albumin-binding paclitaxel (each cycle is 21 days).
  Differences in peripheral neurotoxicity questionaire scores between dominant hands and non-dominant hands after 4 cycles of albumin-binding paclitaxel monotherapy.
Safety of compression gloves in preventing albumin-binding paclitaxel induced neurotoxicity. | From date of consent to one months after Cycle 4 administration of albumin-binding paclitaxel (each cycle is 21 days).
  Adverse events related to compression gloves intervention are collected.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, PhD, Principal Investigator — Department of medical oncology, Fudan University Shanghai Cancer Center
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No